CLINICAL TRIAL: NCT01722773
Title: Trial of Non-invasive Ventilation for Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Lakshmi Durairaj, Staff Physician, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPPV
Record Dates: First submitted 2012-11-01; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipap (Active Comparator): Bipap
  Interventions: Device: Bipap (Respironics, Inc)
- Standard of care (No Intervention): No intervention

INTERVENTIONS:
Device: Bipap (Respironics, Inc) — Bipap every night pressure at 15/5 with heated humidifier
  Other Names: Non-invasive Positive pressure ventilation
  Arms: Bipap

SUMMARY:
The use of domiciliary non-invasive positive pressure ventilation (NPPV) in stable chronic obstructive pulmonary disease (COPD) with chronic hypercapnic respiratory failure has yielded variable effects on survival, quality of life and dyspnea. The investigators hypothesized that use of NPPV in stable COPD might result in improvement in quality of life and dyspnea.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is associated with progressive decline in lung function with resultant chronic respiratory failure. This leads to significant rates of hospitalization, disability, and death. COPD is also associated with sleep disordered breathing and nocturnal hypoventilation, resulting in nocturnal and daytime hypoxemia and hypercapnia. These, in turn, can contribute to fatigue, dyspnea and impaired quality of life. Presence of hypercapnia is associated with a 33% 5-year survival. Nocturnal NPPV can theoretically rest overloaded respiratory muscles, prevent nocturnal hypoventilation, and reset central respiratory drive in patients with hypercapnia. The use of non-invasive positive pressure ventilation (NPPV) in late stage COPD appears logical to change this inexorable course, to alleviate symptoms and to improve quality of life. While NPPV has a definite role in the management of acute hypercapnic respiratory failure, its role in the management of late stage stable COPD is controversial. Multiple studies have shown no survival benefit for nocturnal NPPV in chronic hypercapnic stable COPD patients. The effects on quality of life and dyspnea scores in such patients have been inconsistent. The variable efficacy might have been due to late administration of the intervention in the course of disease, in the presence of advanced hypercapnic respiratory failure. We sought to assess the effect of applying NPPV on indices of health-related quality of life in patients with relative normocapnia. We hypothesized that patients with stable severe COPD have improved quality of life and reduced dyspnea with the use of NPPV.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic obstructive pulmonary disease (COPD) defined as forced expiratory volume in the first second (FEV1)/forced vital capacity (FVC) ratio of <0.70, with at least 10 pack-years smoking history

Exclusion Criteria:

* congestive heart failure, obstructive sleep apnea, chronic respiratory conditions other than COPD, age < 35 years, any disease limiting life expectancy to less than two years, active malignancy other than non-melanotic skin cancer in the previous two years, and with any anatomic variation or disease process that precluded wearing a nasal mask

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
CRDQ | 6 months
  Chronic Respiratory Disease Questionnaire

SECONDARY OUTCOMES:
6-minutes walk test | 6 months
  Walking distances in feet
TDI | 6 months
  Transitional Dyspnea Index
PO2 | 6 months
  Oxygenation
NIF | 6 months
  Negative Inspiratory force

OTHER OUTCOMES:
Side effect questionnaire | 6 months
  Side effects with mask use

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of IOwa, Iowa City, Iowa, United States